CLINICAL TRIAL: NCT06075667
Title: Efficacy, Safety, and Pharmacokinetics of Tirzepatide Once Weekly Versus Placebo in Adolescent Participants Who Have Obesity, or Are Overweight With Weight-Related Comorbidities: A Randomized, Double-Blind Trial (SURMOUNT-ADOLESCENTS)
Brief Title: A Study of Tirzepatide (LY3298176) Once Weekly in Adolescent Participants Who Have Obesity or Overweight With Weight-Related Comorbidities
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17365; I8F-MC-GPHP (Other: Eli Lilly and Company); 2023-504413-80-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants will receive tirzepatide subcutaneously (SC).
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of tirzepatide in adolescents that have obesity or overweight with at least one weight-related comorbidity. The study will last approximately 90 weeks and may include up to 25 visits.

Participants who have completed the primary 72-week GPHP study and have been off treatment for no more than 12 weeks (including the 4-week safety follow-up period), will have the opportunity to receive an additional 156 weeks of treatment with tirzepatide as well as continuing the lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have obesity, as defined by BMI equal to or above the 95th percentile for age and sex, on age- and sex-specific growth chart, OR
* Have overweight, as defined by BMI equal to or above the 85th percentile but less than the 95th percentile for age and sex, on age- and sex-specific growth chart, with at least 1 weight-related comorbidity.

  * dyslipidemia
  * pre-hypertension
  * hypertension
  * nonalcoholic fatty liver disease
  * obstructive sleep apnea
  * prediabetes
  * documented preexisting condition of Type 2 Diabetes

Participants with Type 2 Diabetes Mellitus (T2DM)

* Have been treated with either diet and exercise alone or stable treatment with metformin for at least 90 days prior to screening and have a HbA1c<9.0%

Exclusion Criteria:

* Have a self-reported, or by parent or legal guardian where applicable, decrease in body weight more than 5 kilogram (kg) (11 lbs.) within 90 days before screening irrespective of medical records.
* Have Type 1 Diabetes
* Have taken within 90 days before screening or intend to start prescribed or over-the-counter medications, or alternative remedies including herbal or nutritional supplements, intended to promote body weight reduction.
* Are prepubertal (Tanner stage 1).
* Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome Type 2
* Have a history of chronic or acute pancreatitis.
* Have undergone or plan to undergo weight reduction procedure during the study, such as, but not limited to

  * gastric bypass
  * sleeve gastrectomy
  * restrictive bariatric surgery, such as Lap-Band gastric banding, or
  * any other procedure intended to result in weight reduction.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Mass Index (BMI) | Baseline, Week 72

SECONDARY OUTCOMES:
Percentage of Participants with ≥5% BMI Reduction | Baseline, Week 72
Change from Baseline in Body Weight | Baseline, Week 72
Change from Baseline in Waist Circumference | Baseline, Week 72
Change in Impact of Weight on Quality of Life (IWQOL)-Kids Physical Comfort Domain Score | Baseline, Week 72
Change from Baseline in Body Weight Percentile based on Sex and Age-specific Growth Charts | Baseline, Week 72
Change from Baseline in Systolic Blood Pressure | Baseline, Week 72
Change from Baseline in Diastolic Blood Pressure | Baseline, Week 72
Percent Change from Baseline in Total Cholesterol | Baseline, Week 72
Change from Baseline in Fasting Glucose | Baseline, Week 72
Change from Baseline in Fasting Insulin | Baseline, Week 72
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) of Tirzepatide | Baseline through Week 72
  AUC is presented as a single average measure of AUC across the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (10):
  - CenExel iResearch, LLC, Decatur, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Barry J. Reiner, MD, LLC, Baltimore, Maryland
  - M Health Fairview - Delaware Clinical Research Unit (DCRU), Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Aventiv Research Inc, Columbus, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Vanderbilt Health One Hundred Oaks, Nashville, Tennessee
- Canada (4):
  - Alberta Diabetes Institute, Edmonton, Alberta
  - The Wharton Medical Clinic Clinical Trials Inc, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
- Czechia (5):
  - ReFit Clinic, Olomouc, Olomoucký kraj
  - Nemocnice AGEL Ostrava - Vitkovice a.s., Ostrava, Ostrava Město
  - Fakultni nemocnice v Motole, Prague, Praha 5
  - Nemocnice Jihlava, Jihlava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Israel (7):
  - Yitzhak Shamir Medical Center, Beer Yaacov, Central District
  - Schneider Children's Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Emek Medical Center, Afula, Northern District
  - Rambam Health Care Campus, Haifa, Northern District
  - Soroka Medical Center, Beersheba, Southern District
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona, Veneto
  - Azienda Ospedaliera Universitaria Di Messina G. Martino, Messina
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
- Poland (3):
  - Instytut Diabetologii, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 SUM, Zabrze, Silesian Voivodeship
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Uniwersyteckie Centrum Pediatrii im. M. Konop -T, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide (LY3298176) Once Weekly in Adolescent Participants Who Have Obesity, or Are Overweight With Weight-Related Comorbidities — https://trials.lilly.com/en-US/trial/427361